CLINICAL TRIAL: NCT04113512
Title: Yoga Nasal Irrigation in the Treatment of Chronic Tension Type Headache: Randomised Waitlist Controlled Trial
Brief Title: Yoga Nasal Irrigation in the Treatment of Chronic Tension Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: University of Rajasthan (Unknown); Yog-Kulam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMP/98672
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Chronic Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Nasal Irrigation Group (Experimental): Saline nasal irrigation using neti pot was practiced.
  Interventions: Other: Jalaneti
- Wait list Control group (No Intervention): Group was given usual pain medication. After trial period, they were offered the intervention.

INTERVENTIONS:
Other: Jalaneti — Sterilised and lukewarm isotonic salt water using neti pot was poured into one nostril, so that it leaves through the other. The procedure is then repeated on the other side, and the nose is dried by bending forward and by rapid yoga breathing
  Arms: Yoga Nasal Irrigation Group

SUMMARY:
To evaluate the effectiveness of Yoga Nasal Irrigation (Jalaneti) on patients with chronic tension-type headache reducing pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of chronic tension type headache as per International Classification of Headache Disorders, 3rd edition (beta version) (ICHD-3 beta criteria)
* Aged 18-60 years;
* Ability of understand and completing the headache dairy;
* Volunteering to the study
* Provide written informed consent.

Exclusion Criteria:

* Not having tension-type headache during the pervious 3 months or having less than 8 episode of tension type headache in serious month.
* Taking any prophylactic headache medication or complementary and alternative medicine in last 3 month;
* Secondary Headaches
* In pregnancy, lactation, or planning to be pregnant in 6 months
* Having nose bleeding disorders or recurrent infections;
* Psychiatric diagnosis or medication history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Headache Frequency | Change from baseline to 6 weeks
  Number of days with headache was assessed using headache diary

SECONDARY OUTCOMES:
Headache severity | Change from baseline to 6 weeks
  Mean pain intensity of tension-type headache measured using Visual Analogue Scale from 0-10, 0 defined as no pain and 10 defined as an unbearable pain
Duration of Headache | Change from baseline to 6 weeks
  Duration of each headache attack (hours per day)
Headache disability | Change from baseline to 6 weeks
  Disability caused by headache was measure using Headache Impact Test (HIT-6).

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Yog-Kulam; Jaydeep Joshi, Study Chair — Yog-Kulam; Placheril John, PhD, Study Chair — University of Rajasthan, India; Shekhar Sharma, Study Director — NMP Medical Research Institute, India
Locations (1):
- Yoga Bhavan, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided